CLINICAL TRIAL: NCT06274216
Title: The Effect of Vitamin D Supplementation on Dental Implant Osseointegration: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Dr. Atif Iqbal, Associate Professor, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4381021ABOS
Record Dates: First submitted 2024-01-18; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Osseointegration Failure of Dental Implant
Keywords: Dental implants; ISQ Value; Osseointegration; Vitamin D
MeSH Terms: interventions — Cholecalciferol; Tocopherols

STUDY DESIGN:
Intervention Model Description: The research commences through a self-administered questionnaire such as age, gender, weight, height, BMI, smoking habits, sun exposure, and employment status.
  Prior to implant surgery, each participant undergoes a blood test to assess their vitamin D levels.
  Detailed records are maintained concerning the anatomical position (molar, pre-molar, canine, and incisor) and implant site (maxilla and mandible) for every participant.
  Group Formation: The participant pool is stratified into two distinct groups - Group A and Group B. This categorization is essential for implementing and comparing different interventions within the study. Group A undergoes a specific intervention wherein they receive a daily oral dose of 5000 IU of vitamin D3 for a duration of 12 weeks. In contrast, Group B receives a placebo.
  Following the intervention period, the implants are allowed to cure adequately
Who Masked: Participant, Care Provider
Masking Description: Groups A and B were created out of all patients who had signed up. Patients in group A received 5000 IU of vitamin D3 orally every day for 12 weeks , whereas patients in group B received a placebo. Patients were blinded to the study medication. The implants were then allowed to cure adequately and submerged for a further three months. Patients were summoned back three months later to un-cover the implant.
  The both groups were compared for the difference of osseo-integration at 3 months, as well as difference of osseo-integration were compared with respect to implant site (maxilla and mandible).
  Additionally, change in vitamin D levels were also assessed pre-operatively and post-operatively at 3 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients in group A received 5000 IU of vitamin D3 orally every day for 12 weeks
  Interventions: Drug: Vitamin D3
- Group B (Active Comparator): Patients in group B received 400mg of vitamin E orally every day for 12 weeks
  Interventions: Drug: Vitamin E 400

INTERVENTIONS:
Drug: Vitamin D3 — 5000 IU of vitamin D3 orally every day for 12 weeks
  Other Names: Sunny-D
  Arms: Group A
Drug: Vitamin E 400 — 400mg of vitamin E orally every day for 12 weeks
  Other Names: Evion
  Arms: Group B

SUMMARY:
Dental implantation is a new technique for the single or more missing tooth replacement. Dental professionals might utilize the findings of this investigation to generate local data and learn more about how vitamin D affects bone metabolism and implant osseo-integration. The long-term success of dental implants would also be enhanced and preserved with the right medical use of vitamin D

DETAILED DESCRIPTION:
Treatment option for replacing lost natural teeth is dental implants. Many factors are essential for the dental implant osse-ointegration, consisting of bone quality and volume, surgical approach and complications and host-associated factors like deficient nutritional status. By influencing bone metabolism, vitamin D, together with calcium, is essential for osseo-integrating implants. The significance of vitamin D supplementation in osseo-integration has received little attention in dental literature; there is little data involving people, and the majority of investigations have used animal models. Due to numerous environmental and dietary factors, international data is not applicable to our population. Latest study shows that 54% of the individuals were vitamin D deficient and 31% had vitamin D insufficiency in Pakistan.(Riaz et al., 2016) As well as Pakistani are less likely to expose to sun due to their full clothing, use of veil and Burqah. This research was therefore assessed the impact of vitamin D supplementation during dental implant osseointegration. In this research, the local data have been generated and dental implants in the presence of vitamin-D supplementation were tested for effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Patients of age 18 to 45 years

* Patients of either gender
* Patients undergoing for dental implant
* Patients with Vitamin-D insufficiency

Exclusion Criteria:

Patients with any bone regenerative therapy prior to dental implants

* Patients with arthritis
* Patients with periodontal disease
* Patients with bleeding disorders
* Patients with poor oral hygiene
* Patients with uncontrolled hypertension and diabetes mellitus
* Patients with severe vitamin D deficiency
* Patients with chronic renal disease
* Patients on proton pump inhibitors
* Pregnant women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Osseo-integration is measured by evaluating the ISQ value (Implant Stability Quotient, ranging from 1-100) | 12 weeks
  It will assess the difference in osseo-integration among patients undergoing dental implant procedures. Osseo-integration is measured by evaluating the ISQ value (Implant Stability Quotient, ranging from 1-100) using radiographic and clinical assessments with Ostell. A higher ISQ value indicates greater stability of the dental implants in the surrounding bone tissue. The assessment is conducted three months post-implantation, following a period of implant curing.

SECONDARY OUTCOMES:
Evaluation of Mean Change in Serum Vitamin D Levels in Dental Implant Patients with and without Vitamin D Supplementation at a Tertiary Care Hospital | 12 weeks
  The secondary outcome in this study is to measure the mean change in serum vitamin D levels in both groups. This involves assessing how the serum vitamin D levels evolve over the course of the study in both the group receiving vitamin D supplementation and the group receiving a placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Afifa Razi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The informed consent process typically outlines the extent to which data will be shared. If participants were not informed about individual data sharing, it may be ethically inappropriate to do so.

REFERENCES:
- [Result] Alsulaimani L, Alqarni A, Almarghlani A, Hassoubah M. The Relationship Between Low Serum Vitamin D Level and Early Dental Implant Failure: A Systematic Review. Cureus. 2022 Jan 15;14(1):e21264. doi: 10.7759/cureus.21264. eCollection 2022 Jan. PMID 35178319
- [Result] Munhoz Pereira T, Alvim-Pereira F, Kaiser Alvim-Pereira CC, Ignacio SA, Machado de Souza C, Trevilatto PC. A complete physical mapping of the vitamin D receptor gene for dental implant loss: A pilot study. Clin Oral Implants Res. 2019 Dec;30(12):1165-1178. doi: 10.1111/clr.13529. Epub 2019 Sep 24. PMID 31461186
- [Result] Tabrizi R, Mohajerani H, Jafari S, Tumer MK. Does the serum level of vitamin D affect marginal bone loss around dental implants? Int J Oral Maxillofac Surg. 2022 Jun;51(6):832-836. doi: 10.1016/j.ijom.2021.11.006. Epub 2021 Dec 3. PMID 34872836
- [Result] Werny JG, Sagheb K, Diaz L, Kammerer PW, Al-Nawas B, Schiegnitz E. Does vitamin D have an effect on osseointegration of dental implants? A systematic review. Int J Implant Dent. 2022 Apr 11;8(1):16. doi: 10.1186/s40729-022-00414-6. PMID 35403929
- [Result] Pourshahidi S, Yousefain M. The Relationship Between Serum Level of Vitamin D3 and Osseointegration Around the Dental Implant. J Oral Implantol. 2021 Feb 1;47(1):88-90. doi: 10.1563/aaid-joi-D-19-00341. PMID 32663271